CLINICAL TRIAL: NCT04382378
Title: Effects of Different Regimen Protocols of NMES in COVID 19 Critically Ill Patients
Brief Title: Effects of NMES in Critically Ill Patients
Acronym: NUMBERNMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Escola Superior de Ciencias da Saude (Other)
Responsible Party: Principal Investigator, Vinicius Zacarias Maldaner da silva, Principal Inverstigator, Escola Superior de Ciencias da Saude
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAP042017
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Mechanical Ventilation Complication; Muscle Weakness Condition; Covid19
Keywords: muscular atrophy; electric stimulation therapy; intensive care units
MeSH Terms: conditions — COVID-19; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will be blinded to randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Group that will receive a standard care from physiotherapy staff not involved in delivering the intervention whenever feasible.
- 50 electrically evoked contractions (Experimental): Group that will receive a standard care from physiotherapy staff plus neuromuscular electrical stimulation with the following parameters: pulsed current; freqeuncy 50Hz; pulse witdh 400 us, current intensity that get level 4/5 of evoked contractions proposed by Segers et al; on/off time and duration of therapy that allow 50 ellectrically evoked contractions with surface electrodes positioned on the quadriceps femoris.
  Interventions: Device: neuromuscular electrical stimulation
- 100 electrically evoked contractions (Experimental): Group that will receive a standard care from physiotherapy staff plus neuromuscular electrical stimulation with the following parameters: pulsed current; freqeuncy 50Hz; pulse witdh 400 us, current intensity that get level 4/5 of evoked contractions proposed by Segers et al; on/off time and duration of therapy that allow 100 ellectrically evoked contractions with surface electrodes positioned on the quadriceps femoris.
  Interventions: Device: neuromuscular electrical stimulation

INTERVENTIONS:
Device: neuromuscular electrical stimulation — application of an electric current through electrodes placed on the skin over the targeted musclesto induce skeletal muscle contractions
  Other Names: NMES; transcutenaous electrical nerve stimulation
  Arms: 100 electrically evoked contractions; 50 electrically evoked contractions

SUMMARY:
Muscle wasting occurred early and rapidly in critically ill patients. Early therapeutic strategies to either maintain muscle structure and function should be encouraged. Neuromuscular electrical stimulation (NMES) is an attractive intervention to maintain muscle mass and strength in critically ill patients during the first week of ICU stay. This study will test the hypothesis that the number of contraction per day evoked by NMES in the first two weeks of illness may influence in muscle wasting, with beneficial effects on the physical and functional status in mechanically ventilated patients.

DETAILED DESCRIPTION:
Patients with prolonged mechanical ventilation require deep sedation and mechanical ventilation, factors predisposing to the development of skeletal muscle wasting and acute muscle atrophy. Strategies to attenuate this process must be used. The neuromuscular electrostimulation (NMES) leads to the application of electrical currents in the skin aiming at muscle contraction, has beneficial effects for the population of critical patients. However, the number of contractions induced by NMES to attenuate the loss of muscle mass in this population is not yet established. This randomized controlled trial with 120 patients that will be randomized to one of the 3 study groups: 100 continuous daily contractions (100Cd), 50 continuous daily contractions (50Cd) and control group. Muscle thickness, NMES-induced strength, and clinical and functional parameters at the time of discharge from the ICU and hospital discharge will be assessed daily. The results of this project will provide an important contribution to the understanding of the mechanisms associated with NMES treatment as a tool to minimize the effects of muscle disuse, as well as providing scientific support for the clinical use of this resource in the treatment in the light of the policies' health system.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Intubated and expected to remain invasively mechanically ventilated the day after tomorrow
* laboratory confirmed COVID-19 (diagnosis of SARS-CoV-2 via reverse transcriptase polymerase chain reaction as per the World Health Organization protocol or by nucleic acid based isothermal amplification)

Exclusion Criteria:

* Dependent for activities of daily living in the month prior to current ICU admission (gait aids are acceptable).
* Documented cognitive impairment.
* Proven or suspected spinal cord injury or other neuromuscular disease that will result in permanent or prolonged weakness (not including ICU acquired weakness)
* Death is deemed inevitable as a result of the current illness and either the patient or treating clinical or substitute decision maker are not committed to full active treatment
* pregnancy
* patients with unstable fractures in the vertebral column and lower limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
cross sectional area of rectus femoris | from baseline to 14 days of therapy
  change of muscle wasting assessed by ultrassonogropahy
echointensity of rectus femoris | from baseline to 14 days of therapy
  change of echointensity of rectus femoris assessed by ultrassonography
muscle strength | from baseline to 14 days of therapy
  change of evoked peak torque of quadriceps femoris assesssed by unvolitional testing

SECONDARY OUTCOMES:
Functional status | from baseline to 14 days of therapy
  Functional status assessed by IMS scale ranged from 0 to 10
ICU acquired weakness | from baseline to 14 days of therapy
  percent of patients that have muscle strength assessed by Medical Research Council Sum-Score (MRC-SS) lower than 48

CONTACTS AND LOCATIONS:
Overall Officials: VINICIUS ZACARIAS MALDANER D SILVA, Principal Investigator — Secretaria de Saúde do Distrito Federal
Locations (1):
- Secretaria de Saúde do Distrito Federal, Brasília, Federal District, Brazil